CLINICAL TRIAL: NCT02527915
Title: The Effects of Mental Health eConsults: A Clinic-level Randomized Trial
Brief Title: Mental Health eConsults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Allina Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1507S76668
Record Dates: First submitted 2015-08-14; First posted 2015-08-19 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Mental Disorders
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mental Health eConsults (Experimental): Primary care clinics that will receive the eConsults intervention at the start of the study.
  Interventions: Other: Mental Health eConsults
- Usual care (Active Comparator): Primary care clinics that will deliver care as usual for nine months, and will receive the eConsults intervention nine months subsequent to the eConsults "intervention" clinics.
  Interventions: Other: Care as usual

INTERVENTIONS:
Other: Mental Health eConsults — Providers in primary care clinics who receive the intervention will be able to use electronic consultations (eConsults) with psychiatrists. If a primary care provider wishes to use eConsults, he/she will enter a specific question about a patient in the electronic medical record system and submit as an eConsult. A psychiatrist will review the question and the patient's record, and send a response back to the primary care provider within one business day.
  Arms: Mental Health eConsults
Other: Care as usual — Providers in primary care clinics will deliver care as usual to their patients.
  Arms: Usual care

SUMMARY:
The purpose of this study is to assess whether electronic consultations between primary care providers and psychiatrists affects mental health services delivered in primary care settings.

DETAILED DESCRIPTION:
This study assesses the effects of electronic consultations (eConsults) between primary care providers and psychiatrists as a way to support the delivery of mental health services in primary care settings. The setting for the study are the primary care clinics of Allina Health.

The study uses a randomized rollout design. Across 45 primary care clinics, half of the clinics will be randomly assigned to receive access to eConsults at the start of the study. The other half of the clinics will provide care-as-usual for nine months, at which point they will also gain access to eConsults. Stratified randomization will be used, with stratification on whether primary care clinics have co-located specialty mental health services.

For primary care clinics that are given access to eConsults, the primary care providers in those clinics will have the option of ordering an eConsult on behalf of their patients, which will include specific questions about a particular patient's care. The request is routed to the service region's psychiatry pool, and the psychiatrists have the option of responding. If they choose to respond, the psychiatrist responds with their recommendations within one business day, and the PCP proceeds with care accordingly. The psychiatrist receives 0.75 work relative value units (wRVUs) for providing this service. All communications for the eConsult are routed through Allina's Epic system. Although patients will not be billed for eConsults over the course of the proposed research, some insurance plans do cover it and evidence of eConsult effectiveness may impel other insurers to cover the service.

The study will have two components. First, the investigators will collect web survey data from the primary care providers to assess how access to eConsults affects providers' perceptions of their support and skill for delivering mental health services to their patients. Second, the investigators will assess the effects of receiving eConsults at the patient level, by using data from the Electronic Medical Record system.

ELIGIBILITY:
Inclusion Criteria:

* For the provider surveys, we will recruit all of the primary care providers who work in Allina's primary care clinics to participate in the surveys
* For the patient-level analysis, we will examine data from all patients seen in Allina's primary care clinics during the study period. We will include children and adults.

Exclusion Criteria:

* We will exclude patients from the patient-level analysis who have opted that their secondary data not be used by Allina for research purposes.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 900000 (Estimated)
Dates: Start 2015-08; Primary Completion 2017-01 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Use of eConsults | Within one day of a primary care clinic visit
  Whether an eConsult was actually ordered in a primary care visit for a mental health issue. Data will be extracted from the electronic medical record system.

SECONDARY OUTCOMES:
Frequency of specialist consultation | Baseline and 6 months
  Primary care providers report how often in the past 6 months they consult with a mental health specialist for help with a patient's mental health issues at the baseline web survey questionnaire and the 6-month followup survey. Survey data will be collected from up to 400 primary care providers.
How easy to consult with specialist | Baseline and 6 months
  Primary care providers report how easy it is in the past 6 months to consult with a mental health specialist for help with a patient's mental health issues at the baseline web survey questionnaire and the 6-month followup survey. Survey data will be collected from up to 400 primary care providers.
Patient contact with a specialist, 1 month | 1-month
  Whether patients see a mental health specialist within a month after a primary care visit. Data will be extracted from the electronic medical record system.
Patient contact with a specialist, 3 months | 3-month
  Whether patients see a mental health specialist within 3 months after a primary care visit. Data will be extracted from the electronic medical record system.
Patient contact with a specialist, 6 months | 6-month
  Whether patients see a mental health specialist within 6 months after a primary care visit. Data will be extracted from the electronic medical record system.
Change in depression symptoms | Baseline office visit to followup within 6 months
  Depressive symptoms, as measured by the PHQ-9 at the office visit and again at a routine PHQ9 measurement within six months.
Total cost of care, 1 month | 1-month
  Total health care spending one month after a primary care visit (including the primary care visit). Data will be extracted from the electronic medical record system.
Total cost of care, 3 month | 3-month
  Total health care spending three months after a primary care visit (including the primary care visit). Data will be extracted from the electronic medical record system.
Total cost of care, 6 month | 6-month
  Total health care spending six months after a primary care visit (including the primary care visit). Data will be extracted from the electronic medical record system.
Providers get needed support for mental health care | Baseline and 6 months
  Providers indicate agreement with whether they have adequate support for delivering five aspects of mental health care at the baseline web survey questionnaire and the 6-month followup survey. Survey data will be collected from up to 400 primary care providers.
Any mental health service use, 2 week | 2-week
  Whether any mental health services (medication, counseling) were used after a primary care visit. Data will be extracted from the electronic medical record system.
Any mental health service use, 1 month | 1-month
  Whether any mental health services (medication, counseling) were used after a primary care visit. Data will be extracted from the electronic medical record system.
Any mental health service use, 3-month | 3-month
  Whether any mental health services (medication, counseling) were used after a primary care visit. Data will be extracted from the electronic medical record system.
Any mental health service use, 6 month | 6-months
  Whether any mental health services (medication, counseling) were used after a primary care visit. Data will be extracted from the electronic medical record system.
Provider-perceived patient access | Baseline and six months
  Providers' perceptions of how quickly their patients are able to access needed specialty mental health services at the baseline web survey questionnaire and the 6-month followup survey. Survey data will be collected from up to 400 primary care providers.

OTHER OUTCOMES:
Emergency department use, 1 month | 1-month
  Whether there was any emergency department use in the months after a primary care visit. Data will be extracted from the electronic medical record system.
Emergency department use, 3 months | 3-month
  Whether there was any emergency department use in the three months after a primary care visit. Data will be extracted from the electronic medical record system.
Psychotropic medication use, 1 month | 1-month
  Whether there was any psychotropic drug prescription and use in the month after a primary care visit. Data will be extracted from the electronic medical record system.
Psychotropic medication use, 3 month | 3-month
  Whether there was any psychotropic drug prescription and use in the three months after a primary care visit. Data will be extracted from the electronic medical record system.
Inpatient use, 1 month | 1-month
  Whether there was any emergency department use in the month after a primary care visit. Data will be extracted from the electronic medical record system.
Inpatient use, 3 month | 3-month
  Whether there was any emergency department use in the three months after a primary care visit. Data will be extracted from the electronic medical record system.
Confidence in depression treatment | Baseline and six months
  Providers are asked about their levels of confidence in five aspects of depression treatment at the baseline web survey questionnaire and the 6-month followup survey. Survey data will be collected from up to 400 primary care providers.
Skill in depression treatment | Baseline and six months
  Providers are asked to assess their skill in four aspects of depression treatment at the baseline web survey questionnaire and the 6-month followup survey. Survey data will be collected from up to 400 primary care providers.

CONTACTS AND LOCATIONS:
Overall Officials: Ezra Golberstein, Ph.D., Principal Investigator — University of Minnesota
Locations (1):
- Allina Health, Minneapolis, Minnesota, United States